CLINICAL TRIAL: NCT05899192
Title: Factors Predicting Outcome of Admitted Pneumonia Patients in Critical Care Unit
Brief Title: Outcome Factors of Pneumonia Patients in Critical Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Hamed Sayed Mohamed, Resident doctor, Assiut University
Other Study IDs: Pneumonia in patients at icu
Record Dates: First submitted 2023-05-16; First posted 2023-06-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia Aggravated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the risk factor that affect pneumonic patients at the critical care unit regarding the history investigation and clinical data

DETAILED DESCRIPTION:
Pneumonia remains a serious illness with important clinical impact . It is defined as acute respiratory tract infection that affect lower respiratory tract ,it is classified as community acquired pneumonia (CAP), hospital acquired pneumonia (HAP) and ventilator associated pneumonia .

In this work we assess the factors that affect the prognosis of critically ill patients with pneumonia regarding the age ,sex ,smoking, other co morbidity as diabetes mellitus, hypertension , liver diseases , kidney diseases, heart diseases and chest diseases, clinical date and investigation .

ELIGIBILITY:
Inclusion Criteria:

* 1- Age above 18 yrs.

  2- Critically ill patients admitted to ICU with clinical manifestations of pneumonia in assuit university hospital

Exclusion Criteria:

* 1- Age below 18 yrs. 2- Patients don't have critical illness 3- Patient who refused to contribute in this study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with age above 18 years and below 80 years old with manifestations of pneumonia
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-11-25 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the risk factor that affect pneumonic patients at the critical cre unit and ICU . | 1 year
  to develop and determine the risk factor that affect critically ill patients with pneumonia and the mortality rate .